CLINICAL TRIAL: NCT05426122
Title: Degree of Digestibility of Barley Rice Proteins
Acronym: Bar-pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 6239222600
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Digestive System
Keywords: Barley rice protein; Digestibility; Protein digestion kinetics

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Barley rice protein (Experimental): Barley rice protein powder presented as a shake
  Interventions: Other: Barley rice protein concentrate shake
- Pea protein (Experimental): Pea protein powder presented as a shake
  Interventions: Other: Pea protein concentrate shake
- Whey protein (Experimental): Whey protein powder presented as a shake
  Interventions: Other: Whey protein concentrate shake

INTERVENTIONS:
Other: Barley rice protein concentrate shake — At one out of three test days barley rice protein concentrate powder will be mixed with water to obtain a shake, representing a 20g protein load.
  Arms: Barley rice protein
Other: Pea protein concentrate shake — At one out of three test days pea protein concentrate powder will be mixed with water to obtain a shake, representing a 20g protein load.
  Arms: Pea protein
Other: Whey protein concentrate shake — At one out of three test days whey protein concentrate powder will be mixed with water to obtain a shake, representing a 20g protein load.
  Arms: Whey protein

SUMMARY:
This study aims to assess the degree of digestibility of barley rice protein and compare this to another sustainable, commercially available protein concentrate (pea protein), and a benchmark whey protein, and to assess the effects on blood glucose and insulin levels.

The study is a randomized, cross-over, double blind, controlled trial. Three different treatments, all representing a 20g protein load, will be evaluated with a washout period of minimum one week between the test days. Blood will be collected via a catheter before and up-to five hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via a short questionnaire during each test day. After each test day gastrointestinal complaints are collected via an online questionnaire.

DETAILED DESCRIPTION:
Barley rice protein is extracted from brewer spent grains (BSG), which is the most voluminous by-product of the brewing industry. Until now, BSG has been mainly used for animal feed or is directly discarded, which is an enormous waste of resources and causes serious environmental pollution. BSG is rich in cellulose and non-cellulosic polysaccharides, lignin, and proteins. The protein fraction of BSG contains a relatively high content of the essential amino acid, lysine, in comparison to other cereal products. Because of its high nutritional content, BSG can be applied in human food products for fortification. The digestion characteristics of barley rice protein are not known, but essential to evaluate their future potential as a sustainable protein source.

The primary objective is to estimate the degree of digestibility of barley rice protein by measuring post-prandial amino acid uptake kinetics, and compare this to pea protein and a benchmark protein (whey).

Secondary objectives are to assess the effects on blood glucose and insulin levels.

The study is a randomized, cross-over, double blind, controlled trial. Three different treatments, all representing a 20g protein load, will be evaluated with a washout period of minimum one week between the test days. Blood will be collected via a catheter before and up-to five hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via a short questionnaire during each test day. After each test day gastrointestinal complaints are collected via an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women;
* Age between 18 and 40 years;
* Body mass index (BMI) between 18.5 and 30 kg/m2 ;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor).

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease),or having a condition or disease that may lead to an impaired immune system;
* History of gastrointestinal surgery or having (serious) gastrointestinal complaints;
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery;
* Kidney dysfunction (self-reported);
* Any use of medication that may suppress the immune system, this will be judged by the medical supervisor;
* Use of medication that may influence the study results, such as gastric acid inhibitors, laxatives, stomach protectors and drugs that can affect intestinal motility, this will be judged by the medical supervisor;
* Anaemia (Hb values <7.5 mmol/L for women and <8.5 mmol/L for men);
* Reported slimming, medically prescribed or other extreme diets;
* Use of protein supplements;
* Not willing to give up blood donation during the study;
* Current smokers;
* Alcohol intake ≥4 glasses of alcoholic beverages per day;
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported);
* Abuse of hard drugs;
* Having food allergies and/or intolerances (e.g. for gluten);
* Not having a general practitioner;
* Participation in another clinical trial at the same time;
* Being an employee of the department Food, Health & Consumer Research of Wageningen Food & Biobased Research.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Change in degree of digestibility | During the intervention period on 3 test days: at baseline and postprandial blood samples will be collected from the cannula at 10 time points (T=0, 30, 45, 60, 90, 120, 150, 180, 240, 300 minutes)
  In order to assess change in the degree of digestibility, we determine 19 free amino acids in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption. Blood amino acids will be determined by the laboratory of Wageningen FBR, according a valid method: AccQ-Tag ultra-derivation kit & HPLC.

SECONDARY OUTCOMES:
Change in plasma glucose levels | During the intervention period on 3 test days: at baseline and postprandial blood samples will be collected from the cannula at 10 time points (T=0, 30, 45, 60, 90, 120, 150, 180, 240, 300 minutes)
  Plasma glucose levels will be determined in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption (hospital laboratory Ziekenhuis Gelderse vallei, Ede, the Netherlands)
Change in plasma insulin levels | During the intervention period on 3 test days: at baseline and postprandial blood samples will be collected from the cannula at 10 time points (T=0, 30, 45, 60, 90, 120, 150, 180, 240, 300 minutes)
  Plasma insulin levels will be determined in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption (hospital laboratory Ziekenhuis Gelderse vallei, Ede, the Netherlands).

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No